CLINICAL TRIAL: NCT04741009
Title: A Pre-market, Open-label Feasibility, Prospective, Single-arm Multicenter Feasibility Investigation of Hearing Performance Using the CI632 in Adults With Low-frequency Residual Hearing.
Brief Title: Perimodiolar Implant Performance in Adults With Low-Frequency Residual Hearing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CAM5776
Record Dates: First submitted 2021-01-06; First posted 2021-02-05 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2024-08

CONDITIONS: Sensorineural Hearing Loss; Low-Frequency Residual Hearing
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CI632 Slim Modiolar Electrode (Experimental)
  Interventions: Device: CI632 Slim Modiolar Electrode

INTERVENTIONS:
Device: CI632 Slim Modiolar Electrode — Cochlear Ltd CI632 cochlear implant with Slim Modiolar Electrode

SUMMARY:
The purpose of the feasibility study is to investigate hearing performance (audiometry and speech perception) using the CI632 in a group of adults (n=15) with low-frequency residual hearing who meet inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years-of-age or older at the time of surgery.
2. Low-frequency threshold at 500 Hz ≤ 50 dB HL and high-frequency pure-tone average (PTA), 2000-8000 Hz ≥ 65 dB HL in the ear to be implanted.
3. Pure-tone average (PTA) (0.5k, 1k, 2k Hz) > 30 dB HL in the contralateral ear.
4. CNC word recognition scores (mean of two lists) ≤ 60% in the ear to be implanted and ≤ 80% in the contralateral ear.
5. English spoken as a primary language.
6. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Individuals greater than or equal to 70 years at the time of surgery.
2. Duration of severe to profound sensorineural hearing loss > 20 years per self-report.
3. Onset of sensorineural hearing loss, for the purpose of this study, prior to 5 years-of-age.
4. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array.
5. Conductive overlay of 15 dB or greater at two or more frequencies, in the range of 250 through 1000 Hz in the ear to be implanted.
6. Hearing loss of neural or central origin.
7. Diagnosis of Auditory Neuropathy.
8. Active middle-ear infection.
9. Medical or psychological conditions that contraindicate undergoing surgery as determined by the Investigator.
10. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the device and/or procedure, as determined by the Investigator.
11. Additional handicaps that would prevent or restrict participation in the audiological evaluations as determined by the Investigator.
12. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
13. Investigator site personnel directly affiliated with this study and/or their immediate family (spouse, parent, child, or sibling).
14. Cochlear employees or employees of a Contract Research Organization (CRO) or contractors engaged by Cochlear for the purposes of this investigation.
15. Currently participating, or has participated in the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
To characterize hearing performance of the CI632 in an adult population under expanded indications for use. | 14 months
  To characterize hearing performance of the CI632 using CNC word recognition in quiet scores with percentage correct words.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Midwest Ear Institute, Kansas City, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.